CLINICAL TRIAL: NCT06535217
Title: Explainable Machine Learning for the Assessment of Donor Grafts in Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: the China Liver Transplant Registry (Unknown)
Responsible Party: Principal Investigator, Zhixing Liang, M.D., Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: ZSSY-2403
Record Dates: First submitted 2024-07-28; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Liver Transplant; Complications
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DGF: patients occured delayed graft function after liver transplantation
  Interventions: Procedure: Liver transplantation
- non-DGF: patients NOT occured delayed graft function after liver transplantation
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — Liver transplantation

SUMMARY:
Clinically, organ evaluation generally performed by the senior surgeons based on their experience and the visual and tactual inspection of the graft during procurement. However, it is proved that transplant surgeons intuition in the evaluation of donor risk and the estimation of steatosis is inconsistent and usually inaccurate. Besides, graft assessment is a dynamic process refer to amount of complex factors, which is considered to be an incredibly complicated relationship that is nonlinear in nature. Unfortunately, the classical statistic techniques in vogue such as multiple regression require the statistical assumption of independent and linear relationships between explanatory and outcome variables, and fail to analyse a large number of variables. We attempted to develop liver graft assessment models by predicting postoperative DGF using several ML techniques. Secondly, the best prediction model was selected by comparing the performance of different AI algorithms and logistic regression. Finally, we sought to explain the decision made by AI algorithms using a visualization algorithm based on the best prediction model, helping clinicians evaluate specific organ and whether to receive that may develop DGF postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years-old
2. Underwent deceased donor liver transplantation

Exclusion Criteria:

1. Underwent living-donor LT;
2. Missing rates of data were more than 80%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent deceased donor liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 5636 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Delayed Graft Function (DGF) | Within 7 days after liver transplantation
  defined as early graft dysfunction without the need for a second liver transplant or death

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No